CLINICAL TRIAL: NCT00337909
Title: Computer-Based Training for Cognitive Enhancement: Classroom Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUT-107-2005
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Aging
Keywords: cognitive enhancement; memory; auditory memory; speech; computerized
MeSH Terms: conditions — Speech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Treatment (Experimental): Computerized Plasticity-Based Adaptive Cognitive Training
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Control (Active Comparator): Educational DVDs
  Interventions: Other: Educational DVDs
- No Contact Control (No Intervention)

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Other Names: BrainHQ; Brain Fitness Program
  Arms: Experimental Treatment
Other: Educational DVDs
  Arms: Active Control

SUMMARY:
The primary objective of this study is to evaluate the design and effectiveness of a computer-based training program on the memory and cognitive abilities of mature individuals undergoing healthy aging.

DETAILED DESCRIPTION:
The purpose of this study is to test the new progressions design of a computer-based training program and to demonstrate the effectiveness of this refined cognitive training regimen on participants' performance on normed neuropsychological measures.

Subjects meeting eligibility criteria and providing written, informed consent will complete 40 one hour sessions of a computer based training program.

ELIGIBILITY:
Inclusion Criteria:

A)Participants must be at least 60 years old B)Participants must have a Mini-Mental State Exam (MMSE) score of 24 or higher to ensure that participants do not meet common criteria for dementia C)Participants must be a native English speaker D)Participants must be able to see well enough to read the consent form E)Participants must be able to hear well enough to understand ordinary spoken conversation when the clinical specialist holds a paper in front of his or her face to prevent the participant from lip-reading.

F)Participants must be willing to commit to the time requirements of the study and not have any scheduled trips or absences for more than 1 week during the training.

Exclusion Criteria:

A)Participants must not be planning to begin cholinesterase inhibitor (AChEI) therapy or to change their dosing levels. Subjects currently using AChEI will be included if they have an established steady dosing history at least one month prior to the study and are expected to continue at the same dosage throughout the study.

B)Participants must not have had a head trauma that caused them to lose consciousness in the past five years and have had no subsequent symptoms.

C)Participants must not have had a stroke within the past year; or have had a stroke that has left them with expressive or receptive language problems.

D)Participants must not have any central nervous system disorder that could contribute to cognitive impairment.

E)Participants must not have a tremor preventing the use of a computer mouse or other pointing device.

F)Participants must not currently be active in another clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of training program.

SECONDARY OUTCOMES:
Evaluation of training effects.

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Mahncke, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

REFERENCES:
- [Result] Mahncke HW, Bronstone A, Merzenich MM. Brain plasticity and functional losses in the aged: scientific bases for a novel intervention. Prog Brain Res. 2006;157:81-109. doi: 10.1016/S0079-6123(06)57006-2. PMID 17046669